CLINICAL TRIAL: NCT06002464
Title: Benefit of Acupuncture Combined to Regional Analgesia for Post Operative Pain Relief After Hysterectomy
Acronym: RAACU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VMEC ANEST 16
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: A single center, open label, prospective randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP (Active Comparator): Post operative analgesia with bilateral continuous erector spinae plane block catheter
  Interventions: Procedure: Bilateral ESP catheter
- ESP ACU (Experimental): Post operative analgesia with bilateral continuous erector spinae plane block catheter combined with daily session of acupuncture
  Interventions: Procedure: Acupuncture; Procedure: Bilateral ESP catheter

INTERVENTIONS:
Procedure: Acupuncture — Patient will have session of 30 minutes of acupuncture every day during 3 days
  Arms: ESP ACU
Procedure: Bilateral ESP catheter — Analgesia by Bilateral Continuous erector spine plane block catheter at T9 level for 2 days

SUMMARY:
Since the 90's, the quality of the post operative pain relief is a main concern in most of the healthcare systems in the world. An efficient pain relief improves the quality of recovery after surgery [Level 1A], reduces the risk of persistent pain [level 1A] and makes the patients satisfied.

Continuous regional anesthesia/analgesia promotes a level 1A in quality of postoperative pain relief, reduction in opioids consumption in opioid sparing/free analgesia programs, time to recover and the reduction of hospital stay. However in the postoperative period, breakthrough pain episodes due to mobilization or activity are not well covered by regional analgesia. Furthermore, after removal of the catheter of regional anesthesia, patients may face an unpleasant rebound pain effect.

At VinMec, the technique of regional anesthesia chosen to provide regional analgesia after hysterectomy is a bilateral erector spinae plane block .

Traditional Medicine relieves pain by non-pharmacological methods, especially by acupuncture which bring positive results. Acupuncture has been proven to provide pain relief according to the mechanism of traditional and modern medicine, safe for patients and with few side effects. The acupunture point formula is used by VinMec Sao Phuong Dong Traditional Medicine Center in conjunction with the department of Anesthesiology and Pain management in VinMec Times City International General Hospital to relieve pain after hysterectomy including: Three Yin Intersection (SP-6), Leg Three Miles (ST-36), Taichong (LR-3), Xuehai (SP-10).

The study is to observe the effect of combining acupuncture with regional anesthesia on pain relief and postoperative recovery in patients undergoing hysterectomy.

There is no published study regarding the effects of combining the 2 techniques above as multimodal approach for post operative analgesia after hysterectomy.

DETAILED DESCRIPTION:
Design A single center, open label, prospective randomized controlled trial to study the benefits of combining acupuncture with bilateral continuous ESPB compared to bilateral ESPB alone in patients scheduled for an hysterectomy .

Patient selection At the pre-anesthetic consultation or performed at least 24h before the surgery.

Enrollment and allocation During the pre-anesthetic consultation, if the patient accepts the proven benefits to have surgery performed under combined general anesthesia and regional anesthesia, the anesthesiologist will offer her to participate in the study comparing these two bundles of care using regional anesthesia.

Patients will be assigned via a random number generator into one of two study groups (1 Or 2) by the physician/nurse who obtained consent which is prescribed in the nurse preparation file.

Surgical technique Elective hysterectomy by laparoscopic or Pfannenstiel incision

GROUP 1: ESPB

The ESPB will be performed after the induction of general anesthesia (Décris ton régime d'anesthésie générale). (Kit epidural for adult Tuohy needle 19 G Catheter 20G, Name company). Once hemodynamically stable, the patient will be placed on right lateral decubitus. Right and left side level of puncture is on transverse process of T8 in cephalo-caudal direction. The tip of the catheter should be on the transverse process of T9.

During the ultrasound-guided procedure, the ESP space was located by injecting dextrose 5% to lift up the fascia of the erector spinae muscles off the transverse process. There should be a visible spread of fluid in both cephalad and caudal directions and demonstration of a breathing sign. The catheter 20G will be inserted into this space under US guidance, visualizing the tip of the catheter on the top of the next transverse process, as described above. The catheter placement will be tested by injecting dextrose 5% and demonstrating a cephalo-caudal spread of the liquid in the inter-fascial plane anterior to the ESP muscle. Induction of ESP block will be done 30 min before incision with ropivacaine 0.5% with loading dose as follows:

Patient height (cm) Volume of LA (mL) LEFT RIGHT 140-149 8 6 150-159 10 8 160-169 12 10 170-180 14 12 >180 16 14

Group 2: ESPB combined to Acupuncture Patient will have ESP bilateral catheter as per group 1

Three hours after the surgery, acupuncture will be performed as per the following protocol:

Acupuncture point formula

1. Three Yin Intersection (SP-6): 3 cun above the the highest point of the ankle bone, one finger's breatdth from the posterior border of the tibia
2. Leg Three Miles (ST-36): 3 cun below the knee crease, and approximately one finger's breadth lateral to the tibial crest. It is located near the anterior shin bone muscle, and in a depression between the the fibula and tibia..
3. Taichong (LR-3): put the foot flat on the floor, on the dorsum of the foot, find the point in a depression distal to the junctions of the 1st and 2nd metatarsal bones.
4. Xuehai (SP-10): on the medial border of the patella, in the middle of vastus medialis and sartorius muscle.

Material Acupuncture needle, diameter = 0.25mm, 4cm long, needle material: SUS 304; manufactured by Van Long Medical Equipment Co., Ltd, Wujiang City, China.

Sessions of Acupuncture The patient lies in supine position, with two legs exposed. Acupuncture for 30 minutes,

* At Day 0 The first session will be 3 hours after arrival time in post operative care unit
* At day 1 2 and 3, 2 sessions per day, at 8 am and 3 pm (acupuncture done before the patient starts to do exercises).

Acupuncture performed on both legs. Order of acupuncture points: Three Yin Intersection (SP-6), Leg Three Miles (ST-36), Taichong (LR-3), Xuehai (SP-10)

Acupuncture performed in 2 steps:

* Step 1: needles puncture through the skin at the acupuncture points quickly and decisively.
* Step 2: When needle depth is about 0.5-1cm, manipulate the needle every 10 minutes counterclockwise. At Taichong (LR-3), manipulate the needle every 10 minutes counter-clockwise

Statistical consideration Statistical analysis The study is a superior comparative trial. Patients scheduled for hysterectomy will be randomized into 2 groups: a group receiving standard of care ESPB and a group receiving ESPB + acupuncture. Comparison between groups done for primary and secondary outcomes.

Sample size Assuming the difference in VAS score between two group is 1, variance of VAS score is 2 and equal between two groups, for 95% CI and power of 80%, 32 participants are needed for each group. Assuming loss of follow-up is 10%, a total of 72 participants (36 for each group) is needed.

Analysis plan For primary outcome (VAS score), t-test will be used for the comparison between group. For secondary outcomes, Mann-Whitney test will be used for continuous outcomes and Fisher's exact test will be used for categorical outcomes. All statistical tests are 2 sided with significant level of 0.05.

All analysis will be done with latest version of R statistical software.

Data collection For the first 3 postoperative days, data will be recorded during routine patient rounds done by the anesthesia team in the ICU and surgical ward. Another set of data will be recorded after one month, during routine patient follow-up.

All data will be retrieved from the patient records except for opioid consumption which will be obtained from the PCA pumps. Opioid consumption will be recalculated to morphine milligram equivalents (MMEs).

For pain evaluation, VAS score will be assessed every 2 hours after extubation for 3 consecutive times, and every 8 hours thereafter. Please see table below.

A dedicated anesthesia nurse trained for data collection will follow the patient and collect the data

V. ETHICS Independent Ethics Committee or Institutional Review Board Approval will be obtained from VinMec ethical committee (IRB) and signed by the IRB/IEC chairman or designee before human participants participate in research studies. Before study onset, the protocol, informed consent, advertisements to be used for the recruitment of study participants, and any other written information regarding this study to be provided to the participant or the participant's legal guardian must be approved by the IRB/IEC. Good Clinical Practice (GCP) will be maintained and will be available for review by the Sponsor or its designee.

The investigator is responsible for providing written summaries of the progress and status of the study and written reports on any changes significantly affecting the conduct of the study or increasing the risk to participants.

The study will be performed in accordance with the ethical principles that originated from the Declaration of Helsinki, ICH GCP, and all applicable regulations.

Participant Information and Consent A written informed consent shall be obtained from each participant before entering the study or performing any unusual or nonroutine procedure that involves risk to the participant.

Before recruitment and enrollment, each prospective participant or his or her legal guardian will be given a full explanation of the study, allowed to read the approved ICF, and allowed to have any questions answered. Once the investigator is assured that the participant/legal guardian understands the implications of participating in the study, the participant/legal guardian will be asked to give consent to participate in the study by signing the ICF. The authorized person obtaining the informed consent will also sign the ICF.

ELIGIBILITY:
Inclusion Criteria:

* female
* elective hysterectomy
* accept ton participate
* signed consent

Exclusion Criteria:

* patient refusal
* allergy to local anesthetics
* complex congenital malformation
* mental deficit
* substance abuse(alcohol, drugs, opioids)
* renal insufficiency

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients listed for hysterectomy
Enrollment: 72 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
quality of pain relief | from end of surgery to 3rd day after the surgery
  the area under the curves the Visual analgesia Scores for pain at rest and pain at mobilization

SECONDARY OUTCOMES:
Opioid consumption | from end of surgery to 3rd day after the surgery
  the total morphine consumption used to reach the desired level of pain control
Quality of recovery | measured on 4th day after surgery
  By using a published score of quality of recovery after anesthesia for surgery, the QOR 15

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Macaire, MD, Principal Investigator — Vinmec Healthcare System
Locations (1):
- Vinmec international hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andreae MH, Andreae DA. Local anaesthetics and regional anaesthesia for preventing chronic pain after surgery. Cochrane Database Syst Rev. 2012 Oct 17;10:CD007105. doi: 10.1002/14651858.CD007105.pub2. PMID 23076930
- [Result] Weinstein EJ, Levene JL, Cohen MS, Andreae DA, Chao JY, Johnson M, Hall CB, Andreae MH. Local anaesthetics and regional anaesthesia versus conventional analgesia for preventing persistent postoperative pain in adults and children. Cochrane Database Syst Rev. 2018 Apr 25;4(4):CD007105. doi: 10.1002/14651858.CD007105.pub3. PMID 29694674
- [Result] Simonnet G, Rivat C. Opioid-induced hyperalgesia: abnormal or normal pain? Neuroreport. 2003 Jan 20;14(1):1-7. doi: 10.1097/00001756-200301200-00001. No abstract available. PMID 12544821
- [Result] Richebe P, Cahana A, Rivat C. Tolerance and opioid-induced hyperalgesia. Is a divorce imminent? Pain. 2012 Aug;153(8):1547-1548. doi: 10.1016/j.pain.2012.05.002. Epub 2012 May 17. No abstract available. PMID 22608577
- [Result] Rivat C, Bollag L, Richebe P. Mechanisms of regional anaesthesia protection against hyperalgesia and pain chronicization. Curr Opin Anaesthesiol. 2013 Oct;26(5):621-5. doi: 10.1097/01.aco.0000432511.08070.de. PMID 23995064
- [Result] Richebe P, Rivat C, Liu SS. Perioperative or postoperative nerve block for preventive analgesia: should we care about the timing of our regional anesthesia? Anesth Analg. 2013 May;116(5):969-970. doi: 10.1213/ANE.0b013e31828843c9. No abstract available. PMID 23606468
- [Result] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Result] Richman JM, Liu SS, Courpas G, Wong R, Rowlingson AJ, McGready J, Cohen SR, Wu CL. Does continuous peripheral nerve block provide superior pain control to opioids? A meta-analysis. Anesth Analg. 2006 Jan;102(1):248-57. doi: 10.1213/01.ANE.0000181289.09675.7D. PMID 16368838
- [Result] van Boekel RLM, Warle MC, Nielen RGC, Vissers KCP, van der Sande R, Bronkhorst EM, Lerou JGC, Steegers MAH. Relationship Between Postoperative Pain and Overall 30-Day Complications in a Broad Surgical Population: An Observational Study. Ann Surg. 2019 May;269(5):856-865. doi: 10.1097/SLA.0000000000002583. PMID 29135493
- [Result] Humble SR, Dalton AJ, Li L. A systematic review of therapeutic interventions to reduce acute and chronic post-surgical pain after amputation, thoracotomy or mastectomy. Eur J Pain. 2015 Apr;19(4):451-65. doi: 10.1002/ejp.567. Epub 2014 Aug 4. PMID 25088289
- [Result] Rivat C, Ballantyne J. The dark side of opioids in pain management: basic science explains clinical observation. Pain Rep. 2016 Sep 8;1(2):e570. doi: 10.1097/PR9.0000000000000570. eCollection 2016 Aug. PMID 29392193
- [Result] Kooij FO, Schlack WS, Preckel B, Hollmann MW. Does regional analgesia for major surgery improve outcome? Focus on epidural analgesia. Anesth Analg. 2014 Sep;119(3):740-744. doi: 10.1213/ANE.0000000000000245. No abstract available. PMID 25137006
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Macaire P, Ho N, Nguyen T, Nguyen B, Vu V, Quach C, Roques V, Capdevila X. Ultrasound-Guided Continuous Thoracic Erector Spinae Plane Block Within an Enhanced Recovery Program Is Associated with Decreased Opioid Consumption and Improved Patient Postoperative Rehabilitation After Open Cardiac Surgery-A Patient-Matched, Controlled Before-and-After Study. J Cardiothorac Vasc Anesth. 2019 Jun;33(6):1659-1667. doi: 10.1053/j.jvca.2018.11.021. Epub 2018 Nov 19. PMID 30665850
- [Result] Macaire P, Ho N, Nguyen V, Phan Van H, Dinh Nguyen Thien K, Bringuier S, Capdevila X. Bilateral ultrasound-guided thoracic erector spinae plane blocks using a programmed intermittent bolus improve opioid-sparing postoperative analgesia in pediatric patients after open cardiac surgery: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2020 Oct;45(10):805-812. doi: 10.1136/rapm-2020-101496. Epub 2020 Aug 19. PMID 32817407
- [Result] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Dore C, Williamson PR, Altman DG, Montgomery A, Lim P, Berlin J, Senn S, Day S, Barbachano Y, Loder E. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. JAMA. 2017 Dec 19;318(23):2337-2343. doi: 10.1001/jama.2017.18556. PMID 29260229
- [Result] Bao C, Wang D, Liu P, Shi Y, Jin X, Wu L, Zeng X, Zhang J, Liu H, Wu H. Effect of Electro-Acupuncture and Moxibustion on Brain Connectivity in Patients with Crohn's Disease: A Resting-State fMRI Study. Front Hum Neurosci. 2017 Nov 17;11:559. doi: 10.3389/fnhum.2017.00559. eCollection 2017. PMID 29204113
- [Result] Silva JR, Silva ML, Prado WA. Analgesia induced by 2- or 100-Hz electroacupuncture in the rat tail-flick test depends on the activation of different descending pain inhibitory mechanisms. J Pain. 2011 Jan;12(1):51-60. doi: 10.1016/j.jpain.2010.04.008. Epub 2010 Jun 16. PMID 20554480
- [Result] Lin JG, Lo MW, Wen YR, Hsieh CL, Tsai SK, Sun WZ. The effect of high and low frequency electroacupuncture in pain after lower abdominal surgery. Pain. 2002 Oct;99(3):509-514. doi: 10.1016/S0304-3959(02)00261-0. PMID 12406527
- [Result] Gordon DB, Dahl JL, Miaskowski C, McCarberg B, Todd KH, Paice JA, Lipman AG, Bookbinder M, Sanders SH, Turk DC, Carr DB. American pain society recommendations for improving the quality of acute and cancer pain management: American Pain Society Quality of Care Task Force. Arch Intern Med. 2005 Jul 25;165(14):1574-80. doi: 10.1001/archinte.165.14.1574. PMID 16043674